CLINICAL TRIAL: NCT03400150
Title: CLINICAL PROTOCOL for the INVESTIGATION Of the BioProtect Balloon Implant™ Balloon System Pivotal Study BP-007
Brief Title: BioProtect Balloon Implant™ Balloon System Pivotal Study BP-007
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioProtect (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BP-007
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a 2:1 ratio (balloon implantation:control)
Who Masked: Participant
Masking Description: Study subjects are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- balloon group (Experimental): Marking + balloon implantation + IMRT
  Interventions: Device: balloon
- Control group (Sham Comparator): Marking + IMRT
  Interventions: Other: Control

INTERVENTIONS:
Device: balloon — balloon implantation
  Arms: balloon group
Other: Control — Control - Marking & IMRT are standard of care for prostate cancer - there is no study-specific intervention
  Arms: Control group

SUMMARY:
The BioProtect Balloon Implant™ System is intended to temporarily position the anterior rectal wall away from the prostate during radiotherapy for prostate cancer and in creating this space it is the intent of the balloon to reduce the radiation dose delivered to the anterior rectum. The balloon composed of a biodegradable material that maintains that space for the entire course of prostate radiotherapy treatment and is completely absorbed by the patient's body over time.

DETAILED DESCRIPTION:
This study will be a prospective, multi-center, randomized, double-arm, single blind, concurrently controlled study to assess the safety and efficacy of the balloon in prostate cancer subjects undergoing radiotherapy by means of intensity modulation radiation therapy (IMRT).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Have been histologically diagnosed with invasive adenocarcinoma of the prostate, at clinical stage T1-T3 (as determined by a biopsy taken within 9 months of the screening visit)
* Be scheduled for radiation therapy (XRT) by means of IMRT

Exclusion Criteria:

* Any prior invasive malignancy (except non-melanomatous skin cancer) unless the subject has been disease free for a minimum of 5 years
* Prior radical prostatectomy
* Prior cryosurgery or radiotherapy for prostate cancer, or other local therapy for prostate cancer
* Prior radiotherapy to the pelvis, including brachytherapy
* History of prior surgery involving the rectum or anus
* Prior surgical procedure involving the peri-rectal and/or peri-prostatic area

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (10):
  - Western Radiation Oncology, Apple Valley, California
  - KSK Medical Center, Irvine, California
  - Advanced Urology Institute, Daytona Beach, Florida
  - Rush University Cancer Center, Chicago, Illinois
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Chesapeake Urology Research Associates, Owings Mills, Maryland
  - Urology Nevada, Reno, Nevada
  - Advanced Radiation Center of New York, Lake Success, New York
  - New York University Langone Health, New York, New York
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
- Israel (2):
  - Assuta Ashdod, Ashdod
  - Rabin Medical Center, Petah Tikva
- Maastro, Maastricht, Netherlands
- Institute of Maria Skłodowska-Oncology Centre, Warsaw, Poland
- CUF Porto Instituto, Porto, Portugal
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Company website — http://www.bioprotect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ProSpace Group: Marking + ProSpace implantation + IMRT
  ProSpace: ProSpace balloon implantation
Period: Overall Study
Arm/Group | ProSpace Group | Control Group
Started | 143 | 79
Completed | 139 | 78
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Balloon Group: Marking + Balloon implantation + IMRT
  Balloon implantation
- Total: Total of all reporting groups
Arm/Group | Balloon Group | Control Group | Total
Number analyzed (Participants) | 143 | 79 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (6.29) | 71.1 (7.16) | 70.5 (6.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 143 | 79 | 222
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 13 | 6 | 19
  White | 120 | 65 | 185
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  Netherlands | 13 | 7 | 20
  United States | 55 | 32 | 87
  Poland | 26 | 13 | 39
  Ireland | 5 | 2 | 7
  Israel | 23 | 15 | 38
  Portugal | 18 | 9 | 27
  United Kingdom | 3 | 1 | 4
Localized prostate cancer [Count of Participants; unit: Participants] | 143 | 79 | 222

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint: Number of Subjects in the Balloon and Control Groups With Rectal, Device or Procedure-related Grade > 1 AEs Within 6 Months of Procedure
Description: Non-inferiority in occurrence of rectal, device or procedure-related Grade > 1 AEs within 6 months of implantation for balloon as compared to control group
Time Frame: Within 6 months from balloon implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Group | Control Group
Number analyzed (Participants) | 139 | 78
Participants | 25 | 18

2. Primary Outcome: Efficacy Endpoint: Number of Subjects in the Balloon Group With Reduction of >25% in Rectal Volume Receiving 70 Gy (rV70)
Description: Observed reduction of at least >25% in rectal volume receiving 70 Gy (rV70) in patients after spacer implantation, with efficacy of the study confirmed if >75% of balloon recipients achieved this degree of dose reduction.
Time Frame: 3 months
Population: The balloon spacer implantation was attempted in 143 subjects. The procedure could not be completed for one subject, resulting in an efficacy endpoint population of 142 balloon subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Group
Number analyzed (Participants) | 142
Participants | 139
Statistical Analysis 1: Comparison: Balloon Group; Test type: Other; p = 0.025, Farrington-Manning

ADVERSE EVENTS:
Time Frame: Events within 6 months from implantation
Description: CTCAE 4.0
Arm/Group | Balloon Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/143 | 0/79
Serious Adverse Events (participants affected / at risk) | 12/143 | 10/79
Other Adverse Events (participants affected / at risk) | 108/143 | 60/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Balloon Group (N=143) | Control Group (N=79)
Acute urinary retention (Renal and urinary disorders) | 0 | 1
Cerebral vascular retention (Vascular disorders) | 1 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Rectal bleeding (Product Issues) | 2 | 0
Rectal wall puncture (Product Issues) | 1 | 0
Other (Investigations) | 10 | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Balloon Group (N=143) | Control Group (N=79)
Burning with urination (Renal and urinary disorders) | 14 | 13
Diarrhea (Gastrointestinal disorders) | 12 | 10
Dysuria (Renal and urinary disorders) | 33 | 16
Erectile dysfunction (General disorders) | 9 | 8
Fatigue (General disorders) | 25 | 8
Hot flashes (Renal and urinary disorders) | 10 | 8
Nocturia (Renal and urinary disorders) | 25 | 11
Urgent, frequent urination (Renal and urinary disorders) | 45 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT03400150/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03400150/SAP_001.pdf